CLINICAL TRIAL: NCT06492044
Title: Evaluation of the Association Between Right Atrial Reservoir Strain Variation and Fluid Responsiveness in Patients With Septic Shock
Acronym: RAS-FR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI2022_843_0104
Record Dates: First submitted 2024-06-18; First posted 2024-07-09 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-06

CONDITIONS: Fluid Responsivness; Right Ventricle
Keywords: Right atrial strain; fluid responsivness; preload; right ventricle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- o Patient with septic shock for less than 48 hours (Experimental)
  Interventions: Other: Transthoracic echocardiography (TTE)

INTERVENTIONS:
Other: Transthoracic echocardiography (TTE) — In this pilot study, all included patients will undergo a TTE before (TTEt0) and after (TTEt1) the PLR maneuver, then before (TTEt2) and after the FC (TTEt3).
  Passive leg raising is PLR. FC is fluid challenge. TTE, PLR and FC are routine care procedures in patient in septic shock. In this study the patient will undergo repeated image acquisition with TTE at different times as part of the study, resulting in a longer TTE procedure. The advantage of TTE is that it is a non-invasive, painless, non-irradiating procedure that can be easily performed at the patient's bedside and has no known side effects to date. TTE is a non-invasive procedure that poses no infectious or psychological risk to the patient. No additional follow-up or telephone contact will be necessary for the study. The study concludes once TTEt3 is completed.

SUMMARY:
Evaluating preload dependence is crucial for managing fluid administration in septic shock patients. To avoid unnecessary fluid administration, it's recommended to use dynamic tests like the passive leg raising (PLR) maneuver or a fluid challenge (FC) to see if a patient's cardiac output will increase after fluid resuscitation. Transthoracic echocardiography (TTE) is preferred for this because it can non-invasively, reliably, and reproducibly measure the increase in cardiac output. A patient is considered a "responder" if their stroke volume (SV) increases by more than 15% after an FC. Two-dimensional (2D) right atrial strain (RAS) is a promising tool for evaluating right atrial function. According to the Frank-Starling law, measuring changes in the RA reservoir strain phase (RASr) can identify acute changes in preload, like those induced by a PLR maneuver or an FC.

The aims of this study are to assess the ability of ∆RASr to identify responders after a fluid challenge (FC) and to evaluate the ability of ∆RASr variation induced by a PLR maneuver to distinguish responders from non-responders to volume expansion.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (>18 years old)
* Patient hospitalized in the Intensive Care Unit at Amiens University Hospital with septic shock for less than 48 hours, defined by the presence of all the following criteria: presence of sepsis, hypotension requiring vasopressors to maintain a mean arterial pressure ≥ 65 mmHg despite adequate prior fluid resuscitation, and blood lactate levels > 2 mmol/l (18 mg/dl).
* Patient requiring fluid resuscitation with crystalloids/colloids
* Patient on invasive mechanical ventilation in assisted-controlled mode.
* Blood pressure monitored via a radial or femoral arterial catheter connected to a MostCareUp (Vygon, France).
* Patient or family informed and non-opposition documented.

Exclusion Criteria:

* Poor echocardiographic image quality preventing RASr assessment
* Patient with a contraindication to the PLR maneuver: severe head trauma or intracranial hypertension
* Patient with a history of pericardiectomy
* Patient with a clinical examination consistent with abdominal compartment syndrome
* Patient with aortic pathology, mitral regurgitation greater than grade 2, tricuspid regurgitation greater than grade 2, mitral stenosis, or intracardiac shunt
* Patient with internal or external atrial/ventricular pacing
* Pregnant woman
* Patient on extracorporeal membrane oxygenation and mechanical circulatory support
* Moribund patient
* Patient with supraventricular or ventricular arrhythmia during echocardiographic measurement series
* Patient on renal replacement therapy during echocardiographic examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2022-10-10 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
∆RASrFC value in echocardiography after a fluid challenge | Baseline
  The ∆RASrFC will be defined as the difference between the RASr measured before the FC (RASrt2) and after the FC (RASrt3). To measure the RASr at different times, an acquisition of an apical four-chamber loop image focused on the right atrium will be performed at t0, t1, t2, and t3. The measurement of ∆RASrFC will be done offline, blinded to the results of ∆SVFC, by a cardiac echography expert using dedicated software.
  T0 : refers to the time before the PLR maneuver
∆RASrFC value in echocardiography after a fluid challenge | 10 minutes
  The ∆RASrFC will be defined as the difference between the RASr measured before the FC (RASrt2) and after the FC (RASrt3). To measure the RASr at different times, an acquisition of an apical four-chamber loop image focused on the right atrium will be performed at t0, t1, t2, and t3. The measurement of ∆RASrFC will be done offline, blinded to the results of ∆SVFC, by a cardiac echography expert using dedicated software.
  T1 refers to the time during the PLR maneuver at the peak of the maximal velocity of the aortic VTI.
∆RASrFC value in echocardiography after a fluid challenge | 30 minutes
  The ∆RASrFC will be defined as the difference between the RASr measured before the FC (RASrt2) and after the FC (RASrt3). To measure the RASr at different times, an acquisition of an apical four-chamber loop image focused on the right atrium will be performed at t0, t1, t2, and t3. The measurement of ∆RASrFC will be done offline, blinded to the results of ∆SVFC, by a cardiac echography expert using dedicated software.
  T2 refers to the time before the fluid challenge (FC)
∆RASrFC value in echocardiography after a fluid challenge | 45 minuntes
  The ∆RASrFC will be defined as the difference between the RASr measured before the FC (RASrt2) and after the FC (RASrt3). To measure the RASr at different times, an acquisition of an apical four-chamber loop image focused on the right atrium will be performed at t0, t1, t2, and t3. The measurement of ∆RASrFC will be done offline, blinded to the results of ∆SVFC, by a cardiac echography expert using dedicated software.
  T3 period refers to the time after the end of the FC (15 minutes).

SECONDARY OUTCOMES:
∆RASr value after the PLR maneuver | 10 minutes
  o ∆RASrPLR will be defined as the difference between the RASr measured before the PLR maneuver (RASrt0) and the RASr measured during the PLR maneuver at the peak of the maximal velocity of the aortic VTI (RASrt1).
  T1 period refers to the time during the PLR maneuver at the peak of the maximal velocity of the aortic VTI.
Comparison between SV measured by TTE and SV measured | 10 minutes
  Comparison between SV measured by TTE and SV measured by MostCareUp during the PLR maneuver and the FC.
  SV measured by MostCareUp is based on the PRAM (pressure recording analytical method). This is an uncalibrated monitoring method based on pulse wave analysis.
  the T1 period refers to the time during the PLR maneuver at the peak of the maximal velocity of the aortic VTI.
Association between RASr and CVP | 45 minutes
  Evaluation of the association between RASr, ∆RASrFC, CVP and ∆CVP. ∆CVPFC will be defined as the difference between the CVP measured at time t2 and at time t3. CVP is measured at end-expiration using a jugular venous catheter and will be the average of three consecutive measurements.
  T3 period refers to the time after the end of the FC
Evaluation of right ventricular-arterial coupling in the context of septic shock | Baseline
  Right ventricular-arterial coupling is measured by TTE at times t0, t1, t2 and t3 using a four-chamber view and the TAPSE/PASP parameter.
Evaluation of right ventricular-arterial coupling in the context of septic shock | 10 minutes
  Right ventricular-arterial coupling is measured by TTE at times t0, t1, t2 and t3 using a four-chamber view and the TAPSE/PASP parameter.
Evaluation of right ventricular-arterial coupling in the context of septic shock | 30 minutes
  Right ventricular-arterial coupling is measured by TTE at times t0, t1, t2 and t3 using a four-chamber view and the TAPSE/PASP parameter.
Evaluation of right ventricular-arterial coupling in the context of septic shock | 45 minutes
  Right ventricular-arterial coupling is measured by TTE at times t0, t1, t2 and t3 using a four-chamber view and the TAPSE/PASP parameter.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, France

IPD SHARING:
Plan to Share IPD: No